CLINICAL TRIAL: NCT01058720
Title: A Pilot Study to Evaluate the Efficacy of Daily Vitamin D3 Supplementation in Normal Weight Adolescents
Brief Title: Efficacy of Daily Vitamin D3 Supplementation in Normal Weight Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Seema Kumar, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-004969
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Supplementation; Adolescence
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin D3 (Experimental): Patients would receive 2000 IU of vitamin D3 daily for 12 weeks
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 2000 IU orally once daily for 12 weeks

SUMMARY:
The study is designed to evaluate the increment of serum 25 (OH) vitamin D levels in normal weight adolescents following a 12-week supplementation with Vitamin D3 2000 IU/day.

DETAILED DESCRIPTION:
Twenty normal weight adolescents between ages 12-18 that are age and gender would receive vitamin D3 supplementation at a dose of 2000 IU/day. Levels of 25(OH)vitamin D would be measured at baseline and after 12 weeks.Relationship between 25 OH vitamin D levels and other demographic variables will be assessed.The primary endpoint in this study is the 25 OH Vitamin D level at 12 weeks.

ELIGIBILITY:
Inclusion criteria:

* Subjects between ages 12 and 18 years with BMI between the 5th and the 85th percentile for age and gender.

Exclusion Criteria:

* Subjects with 25 (OH)- D levels >80 ng/mL
* Serum calcium >10.8 mg/dL
* Serum phosphorus > 5.5 mg/dl
* Pregnancy or nursing
* Current cancer
* Patients on multivitamin supplementation
* Dietary calcium intake exceeding 1500 mg/day
* Hepatic or renal disorders
* Type 1 or Type 2 diabetes mellitus
* Those receiving insulin, metformin, or oral hypoglycemic medications
* Malabsorption disorders (Celiac disease, Cystic fibrosis, Inflammatory bowel disease)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Increment in 25(OH)vitamin D level | 12 weeks

SECONDARY OUTCOMES:
Serum Calcium | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seema Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States